CLINICAL TRIAL: NCT01391273
Title: A Multicenter, Double-masked, Randomized, Parallel-group Study Assessing the Safety and Efficacy of Once-Daily Application of Bimatoprost Solution 0.03% Compared to Vehicle in Increasing Overall Eyelash Prominence in Japanese Subjects With Hypotrichosis of the Eyelashes
Brief Title: Safety and Efficacy Study of Bimatoprost in Japanese Patients With Eyelash Hypotrichosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-059
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Eyelash Hypotrichosis
MeSH Terms: interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bimatoprost solution 0.03% (Experimental): One drop of bimatoprost solution 0.03% applied along each upper eyelid margin once daily in the evening for 4 months.
  Interventions: Drug: bimatoprost solution 0.03%
- bimatoprost vehicle solution (Placebo Comparator): One drop of bimatoprost vehicle solution applied along each upper eyelid margin once daily in the evening for 4 months.
  Interventions: Drug: bimatoprost vehicle solution

INTERVENTIONS:
Drug: bimatoprost solution 0.03% — One drop of bimatoprost solution 0.03% applied along each upper eyelid margin once daily in the evening for 4 months.
  Other Names: LATISSE®
  Arms: bimatoprost solution 0.03%
Drug: bimatoprost vehicle solution — One drop of bimatoprost vehicle solution applied along each upper eyelid margin once daily in the evening for 4 months.
  Arms: bimatoprost vehicle solution

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost solution 0.03% compared with vehicle in Japanese adults with hypotrichosis of the eyelashes.

ELIGIBILITY:
Inclusion Criteria:

* Have inadequate eyelashes

Exclusion Criteria:

* Any disease/infection/abnormality of the eye or area around the eye
* Any ocular surgery within 3 months or anticipated need for ocular surgery during the study
* Any permanent eyeliner or implants of any kind or anticipated use of false eyelashes
* Any semi-permanent eyelash tint, dye, curl or eyelash extension application within 3 months
* Use of any over-the-counter eyelash growth product within 6 months or any use of prescription eyelash growth products
* Use of treatments which may affect hair growth (eg, minoxidil, chemotherapy) within 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2012-05-19 (Actual); Study Completion 2012-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Background] Harii K, Arase S, Tsuboi R, Weng E, Daniels S, VanDenburgh A. Bimatoprost for eyelash growth in Japanese subjects: two multicenter controlled studies. Aesthetic Plast Surg. 2014 Apr;38(2):451-60. doi: 10.1007/s00266-014-0293-7. Epub 2014 Mar 19. PMID 24643895

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Started | 88 | 85
Completed | 84 | 83
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution | Total
Number analyzed (Participants) | 88 | 85 | 173
Age, Customized [Number; unit: Participants]
  < 45 Years | 58 | 48 | 106
  45 to 65 Years | 29 | 37 | 66
  >65 Years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 76 | 155
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1-Grade Increase in Overall Eyelash Prominence Using the Global Eyelash Assessment Scale (GEA)
Description: The investigator evaluated the patient's eyelash prominence using the GEA 4-point scale: 1= minimal, 2= moderate, 3= marked and 4= very marked at Baseline and Month 4. At least a 1-grade increase in the GEA score from Baseline indicated improvement.
Time Frame: Baseline, Month 4
Population: Intent to treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 88 | 85
Percentage of participants | 77.3 | 17.6

2. Secondary Outcome: Change From Baseline in Eyelash Length as Measured by Digital Image Analysis (DIA)
Description: Photographs were taken of the eyelashes and assessed using DIA. Length was measured in millimeters (mm). Data from both eyes were averaged for each participant for analysis. A positive change from Baseline indicated longer length (improvement).
Time Frame: Baseline, Month 4
Population: Intent to treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 88 | 85
mm
  Baseline | 6.92 (0.810) | 7.00 (0.825)
  Change from Baseline at Month 4 | 1.62 (1.114) | -0.04 (0.362)

3. Secondary Outcome: Change From Baseline in Eyelash Thickness as Measured by DIA
Description: Photographs were taken of the eyelashes and assessed using DIA. Eyelash thickness (fullness) was assessed across both eyes as an average and is measured in millimeters squared (mm^2). A positive change from Baseline indicated fuller eyelashes (improvement).
Time Frame: Baseline, Month 4
Population: Participants from the Intent to treat population with data available for analysis.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 88 | 84
mm^2
  Baseline | 0.98 (0.318) | 1.01 (0.327)
  Change from Baseline at Month 4 | 0.35 (0.306) | -0.03 (0.195)

4. Secondary Outcome: Change From Baseline in Eyelash Darkness as Measured by DIA
Description: Photographs were taken of the eyelashes and assessed using DIA. Eyelash darkness was measured in both eyes and averaged for analysis using a scale where 0=black and 255=white. A negative change from Baseline indicated darker eyelashes (improvement).
Time Frame: Baseline, Month 4
Population: Participants from the Intent to treat population with data available for analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 88 | 84
Units on a scale
  Baseline | 147.57 (20.340) | 145.27 (18.069)
  Change from Baseline at Month 4 | -12.02 (10.967) | 1.38 (10.854)

ADVERSE EVENTS:
Description: The safety population (all randomized and treated participants) was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Serious Adverse Events (participants affected / at risk) | 2/87 | 2/85
Other Adverse Events (participants affected / at risk) | 12/87 | 6/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Solution 0.03% (N=87) | Bimatoprost Vehicle Solution (N=85)
Appendicitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Solution 0.03% (N=87) | Bimatoprost Vehicle Solution (N=85)
Nasopharyngitis (Infections and infestations) | 12 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.